CLINICAL TRIAL: NCT00788112
Title: A Window Trial of Vorinostat in Patients With Ductal Carcinoma in Situ (DCIS) of the Breast
Brief Title: Vorinostat in Treating Women With Ductal Carcinoma in Situ of the Breast
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: University of California, San Francisco (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: CDR0000617655; UCSF-077532; H10367-31833; UCSF-07031833
Record Dates: First submitted 2008-11-07; First posted 2008-11-10 (Estimated); Last update posted 2017-08-07 (Actual); Status verified 2017-08

CONDITIONS: Breast Cancer
Keywords: ductal breast carcinoma in situ
MeSH Terms: conditions — Breast Neoplasms; Carcinoma, Intraductal, Noninfiltrating | interventions — Vorinostat; Immunohistochemistry; Neoadjuvant Therapy

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Vorinostat (Experimental)
  Interventions: Drug: vorinostat; Genetic: protein expression analysis; Other: immunohistochemistry staining method; Other: laboratory biomarker analysis; Procedure: neoadjuvant therapy; Procedure: therapeutic conventional surgery

INTERVENTIONS:
Drug: vorinostat
Genetic: protein expression analysis
Other: immunohistochemistry staining method
Other: laboratory biomarker analysis
Procedure: neoadjuvant therapy
Procedure: therapeutic conventional surgery

SUMMARY:
RATIONALE: Vorinostat may stop the growth of tumor cells by blocking some of the enzymes needed for cell growth.

PURPOSE: This clinical trial is studying how well vorinostat works in treating women with ductal carcinoma in situ of the breast.

DETAILED DESCRIPTION:
OBJECTIVES:

* To evaluate the in vivo molecular and biological effects of vorinostat by analyzing changes in proliferation and apoptosis, histone acetylation, and HDAC protein expression in women with ductal carcinoma in situ of the breast.

OUTLINE: Patients receive oral vorinostat twice a day for 3 days in the absence of unacceptable toxicity. Patients then undergo lumpectomy or mastectomy 2 hours after the last dose of vorinostat.

Blood and tissue samples are collected at baseline and during surgery for biomarker laboratory studies. Samples are analyzed by immunohistochemistry for Ki-67, HDAC1 and HDAC6 protein expression, and histone H4 and α-tubulin acetylation.

After completion of study therapy, patients are followed for 1 month and then every 6 months for 5 years.

ELIGIBILITY:
DISEASE CHARACTERISTICS:

* Histologically confirmed (by core biopsy) ductal carcinoma in situ

  * Stage 0 disease
* Hormone receptor status not specified

PATIENT CHARACTERISTICS:

* Menopausal status not specified
* ECOG performance status 0-2
* ANC ≥ 1,500/mm^3
* Platelet count ≥ 100,000/mm^3
* Hemoglobin ≥ 9 g/dL
* Potassium and magnesium levels normal
* Prothrombin time or INR ≤ 1.5 times upper limit of normal (ULN) (unless the patient is receiving therapeutic anticoagulation)
* Partial thromboplastin time ≤ 1.2 times ULN (unless the patient is receiving therapeutic anticoagulation)
* Serum creatinine ≤ 1.5 times ULN OR creatinine clearance ≥ 60 mL/min
* Not pregnant or nursing
* Negative pregnancy test
* Fertile patients must use 2 effective barrier methods of contraception
* No known psychiatric or substance abuse disorder that would preclude cooperation with the study requirements
* No active hepatitis A, B, or C infection
* No active HIV infection
* No other active infection
* No other malignancy within the past 5 years
* No condition that would interfere with the absorption or intake of vorinostat
* No history or current evidence of any condition or laboratory abnormality that would confound study results, interfere with the patient's participation in the full duration of the study, or that would not be in the best interest of the patient to participate

PRIOR CONCURRENT THERAPY:

* More than 2 weeks since prior IV antibiotics, antivirals, or antifungals
* No prior gastrointestinal surgery or other procedure that would interfere with the absorption or intake of vorinostat
* No prior or concurrent therapy with any other HDAC inhibitor, including valproic acid
* No prior treatment with any other investigational agent
* No concurrent systemic steroids
* No concurrent anticancer chemotherapy, radiotherapy, biological therapy, or other investigational therapy

Ages: 18 Years to 120 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 17 (Actual)
Dates: Start 2009-07; Primary Completion 2011-11-03 (Actual); Study Completion 2015-08-11 (Actual)

PRIMARY OUTCOMES:
Reduction in Ki-67 compared to baseline Ki-67 | 3 days prior to surgery

SECONDARY OUTCOMES:
Changes in HDAC1 and HDAC6 expression and histone H4 and α-tubulin acetylation in breast tissue and serum samples | 3 days prior to surgery

CONTACTS AND LOCATIONS:
Overall Officials: Laura Esserman, MD, MBA, Principal Investigator — University of California, San Francisco
Locations (1):
- UCSF Helen Diller Family Comprehensive Cancer Center, San Francisco, California, United States